CLINICAL TRIAL: NCT06905964
Title: Effects of Eccentric Cycling Exercise Training With Assistive Devices on Phenotypes and Mitochondrial Metabolism in T Lymphocytes in Sedentary Men
Brief Title: Eccentric Cycling Exercise With Assistive Devices on Mitochondrial Metabolism in T Lymphocyte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202202314A3
Record Dates: First submitted 2025-01-08; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: There Are no Conditions Under Study. Healthy Volunteers
Keywords: Eccentric cycling exercise; Neuromuscular electrical stimulation; Compressive garment; Lymphocyte; Mitochondria
MeSH Terms: interventions — Self-Help Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Eccentric cycling exercise (ECC) (Experimental): High intensity cycling training from 80% to 120% Wmax in eccentric type
  Interventions: Behavioral: Eccentric cycling exercise (ECC)
- Eccentric cycling exercise with assistive devices (ECA) (Experimental): High intensity cycling training from 80% to 120% Wmax in eccentric type (intensity matched the ECC)
  Interventions: Behavioral: Eccentric cycling exercise with assistive devices (ECA)
- Control group (No Intervention): Perform no exercise training but maintain only regular daily lives only in the study.

INTERVENTIONS:
Behavioral: Eccentric cycling exercise (ECC) — Performed exercise training 5 days a week for 5 weeks on an eccentric ergometer.
  Each training session: 5 min at 30% of maximal workload (Wmax) for warmed up and cold down and 30 min the main training phase.
  After each training session, rest in sitting position for 20 min. Exercise intensity: Firstly, set at 80% Wmax, and progressively increased 5% per week to 120 % Wmax in the last week.
  Arms: Eccentric cycling exercise (ECC)
Behavioral: Eccentric cycling exercise with assistive devices (ECA) — Performed exercise training 5 days a week for 5 weeks on an eccentric ergometer.
  Each training session: 5 min at 30% of maximal workload (Wmax) for warmed up and cold down and 30 min the main training phase.
  After each training session, receive NMES in sitting position for 20 min.
  Intensity: Firstly, set at 80% Wmax, and progressively increased 5% per week to 120 % Wmax in the last week.
  Arms: Eccentric cycling exercise with assistive devices (ECA)

SUMMARY:
Eccentric cycling exercise can be a promising modality fwith lower respiratory demands and higher power output. Assistive devices like neuromuscular electrical stimulation (NMES) and compressive garment (CG) accelerates muscle pumping and relieve the eccentric exercise-induced muscle soreness.

Phenotypes and mitochondrial metabolism are crucial to regulate acquired immnunity of T lymphocytes. The study aimed to investigate the effects of eccentric cycling exercise training combined with NMES and CG on mitochondrial phenotypes and bioenergetics in T lymphocytes in sedentary males. The hypothesis were an acute/intense exercise decreased the mitochondrial respiratory capacities of OXPHOS, ETS and bioenergetics, while eccentric cycling training could elevate the diminished mitochondrial functions.

Methods: Twelve sedentary healthy males were randomly assigned to either eccentric cycling with assistive devices (ECA, n=10) or eccentric cycling only (ECC, n=10). All participants performed ECA or ECC at an intensity of 60% to 120% maximal workload progressively on a costumed bicycle ergometer for 40 min/day, 5 days/week for 5 weeks. ECA performed NMES for 20min/session after cycling, while ECC was seated for resting 20 min. Systemic aerobic fitness, phenotypes of T lymphocytes, mitochondrial OXPHOS, ETS respiratory capacities, and bioenergetics in T lymphocytes were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle (exercise<20min/session; <1session/week for a year or longer).
* Nonsmokers, nonusers of medications/vitamins.
* No any cardiopulmonary, neuromuscular, and hematological risks.

Exclusion Criteria:

* Have regular exercise habits (i.e., exercise frequency once per week, duration >20 min).
* Have retabolic or musculoskeletal disease.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to the blood experiments, we recruited male participants only to avoid interference of menstrual cycle.
Enrollment: 30 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mitochondrial bioenergetics of oxygen consumption rate in T lymphocyte | At baseline and 2 days after completing the 5-week intervention
  The bioenergetic health index (BHI) of mitochindria in T lymphocyte was measured. BHI is a parameter for detecting the health status of mitochondrial and efficiency of energy metabolism.
Systemic aerobic fitness (VO2) | At baseline and 2 days after completing the 5-week intervention
  VO2max was determined during the exercise testing. VO2max is the maximum of oxygen deliver and utilization.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Guishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YC, Cheng ML, Tang HY, Huang CY, Chen KM, Wang JS. Eccentric Cycling Training Improves Erythrocyte Antioxidant and Oxygen Releasing Capacity Associated with Enhanced Anaerobic Glycolysis and Intracellular Acidosis. Antioxidants (Basel). 2021 Feb 13;10(2):285. doi: 10.3390/antiox10020285. PMID 33668606
- [Background] Peng SC, Lin YT, Hsu CC, Fu TC, Wang JS. Effects of concentric and eccentric exercise regimens on bioenergetic efficiency of lymphocytes in sedentary males. Eur J Sport Sci. 2024 Dec;24(12):1830-1843. doi: 10.1002/ejsc.12221. Epub 2024 Nov 9. PMID 39520384
- [Background] Huang YC, Hsu CC, Fu TC, Wang JS. Interval aerobic/resistance exercise training depresses adrenergic-induced apoptosis of lymphocytes in sedentary males. Eur J Appl Physiol. 2024 Mar;124(3):837-848. doi: 10.1007/s00421-023-05311-3. Epub 2023 Sep 15. PMID 37712975